CLINICAL TRIAL: NCT02947438
Title: A Prospective, Randomized, Double Blind, Parallel Group Study to Evaluate a 1:1 Dose Conversion From EPREX to EPIAO in Term of Clinical Efficacy and Safety in Subjects With End-Stage Renal Disease on Haemodialysis
Brief Title: Biosimilar Erythropoietin in Anaemia Treatment (Maintenance Phase Study)
Acronym: BEAT_002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Collaborators: Navitas Life Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSS_EP_002
Record Dates: First submitted 2016-10-26; First posted 2016-10-27 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-03

CONDITIONS: Renal Anemia
Keywords: Renal anemia; Haemodialysis; Maintenance phase
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference group (Active Comparator): Generic name: recombinant human erythropoetin injection which is indicated for the treatment of anaemia caused by chronic renal disease.
  Dosage form:Injection Strength: 2000IU, 3000IU, 4000IU
  Frequency and Dosage: Intravenously injection 1-3 times a week for a period of 52 weeks.
  Interventions: Drug: EPREX®
- Experimental group (Experimental): Generic name: recombinant human erythropoetin injection which is indicated for the treatment of anaemia caused by chronic renal disease.
  Dosage form: Injection Strength: 2000IU, 3000IU, 4000IU
  Frequency and Dosage: Intravenously injection 1-3 times a week for a period of 52 weeks.
  Interventions: Drug: EPIAO®

INTERVENTIONS:
Drug: EPREX® — Recombinant human erythropoietin falls under the pharmacological class of haematopoietic / anti anaemic agents. It has been developed for the treatment of anaemia in subjects with chronic kidney disease.
  Erythropoietin, also known as EPO, is a glycoprotein hormone that controls erythropoiesis, or RBC production. It is a cytokine (protein signalling molecule) for erythrocyte precursors in the bone marrow. Human EPO has a molecular weight of 34,000.
  Other Names: Recombinant human erythropoietin
  Arms: Reference group
Drug: EPIAO® — Recombinant human erythropoietin falls under the pharmacological class of haematopoietic / anti anaemic agents. It has been developed for the treatment of anaemia in subjects with chronic kidney disease.
  Erythropoietin, also known as EPO, is a glycoprotein hormone that controls erythropoiesis, or RBC production. It is a cytokine (protein signalling molecule) for erythrocyte precursors in the bone marrow. Human EPO has a molecular weight of 34,000.
  Other Names: Recombinant human erythropoietin
  Arms: Experimental group

SUMMARY:
This study is aimed to comprehensively establish the bio-similarity/bioequivalence in EPIAO® and EPREX® in terms of 52-week comparisons in efficacy, safety and immunogenicity. The targeted population is anaemia patients with end-stage chronic renal disease who previously received epoetin treatment and on haemodialysis.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind, parallel group two arm study to establish the therapeutic equivalence, safety and tolerability of EPIAO® as compared to EPREX® in the treatment of CKD related anaemia in subjects who are on haemodialysis. A total of 264 subjects will be randomized into two groups in a 1:1 ratio. Treatment arm A will receive EPIAO® 1-3 times a week, intravenously for period of 52 weeks and treatment arm B will receive EPREX, 1-3 times a week, intravenously for period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the age of 18 to 75 years
* Subjects with end stage renal disease (CKD stage 5) on hemodialysis and on epoetin treatment for at least 3 months prior to screening
* Subjects with haemoglobin between 10 g/dl to 12 g/dl
* Subjects who are on clinically stable haemodialysis (defined as no clinically relevant changes of dialysis regimen and/or dialyzer) for at least 3 months prior to screening
* Subjects willing to provide a written informed consent
* Subjects with serum ferritin ≥ 200 μg/L and/or transferrin saturation ≥ 20%
* Subjects with a life expectancy of more than at least study period in clinical judgment of the investigator

Exclusion Criteria:

* Subjects with anaemia due to other reasons (that is not renal anaemia)
* Subjects who have undergone blood transfusion within the last 3 months
* Subjects with major complication such as severe/chronic infections or bleeding or aluminum toxicity
* Subjects with suspected or known pure red cell aplasia (PRCA)
* Subjects with a history of aplastic anaemia
* Subjects with uncontrolled diabetes (fasting blood glucose > 240 mg/dl) or uncontrolled hypertension (systolic blood pressure > 180 mm Hg, diastolic blood pressure > 110 mm Hg)
* Subjects with known hypersensitivity to any of the ingredients of the investigational products, the mammalian cell-derived product or human albumin products
* Subjects with history of seizure disorder
* Subjects with hematological disorder
* Subjects with hyperparathyroidism
* Subjects with congestive heart failure and/or angina (NYHA class III and IV)
* Subjects with myocardial infarction or stroke in the preceding 6 months of screening
* Subjects with active malignancy in the previous 5 years
* Subjects with gastrointestinal bleeding in the past 6 months
* Subjects with immunosuppressive therapy in the previous 3 months
* Subjects with active hepatitis B virus (HBsAg) (positive for HBsAg and IgM anti-HBc) and hepatitis C virus (HCV) (positive for Anti-HCV antibody) and human immunodeficiency virus (HIV)
* Female subjects who are pregnant, breast-feeding, planning to be pregnant during the study, or women of child-bearing potential (any woman who is not surgically sterile i.e. bilateral tubal ligation, total hysterectomy or < 2 years post menopause) not using a reliable method of double contraception (e.g. condom plus diaphragm, condom or diaphragm plus spermicidal gel/foam, tubal ligation, or stable dose of hormonal contraception) throughout the study period
* Subjects participating in trials involving erythropoietin in the past 6 months before screening.Subjects currently participating or participation in an investigational study within 30 days prior screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2015-12; Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

PRIMARY OUTCOMES:
Mean absolute change in haemoglobin level from baseline to 6 months | from baseline to 6 months
  Mean absolute change in haemoglobin level from baseline to 6 months after treatment with EPIAO/EPREX in parallel groups (g/dl).
Mean absolute change in weekly epoetin dosage per kg body weight from baseline to 6 months | from baseline to 6 months
  Mean absolute change in weekly epoetin dosage per kg body weight from baseline to 6 months after treatment with EPIAO/EPREX in parallel groups (IU/kg/week).

SECONDARY OUTCOMES:
Mean absolute change in haemoglobin level from baseline to 9 months | from baseline to 9 months
  Mean absolute change in haemoglobin level from baseline to 9 months after treatment with EPIAO/EPREX in parallel groups (g/dl).
Mean absolute change in weekly epoetin dosage per kg body weight from baseline to 9 months | from baseline to 9 months
  Mean absolute change in weekly epoetin dosage per kg body weight from baseline to 9 months after treatment with EPIAO/EPREX in parallel groups (IU/kg/week).
Proportion of subjects with hemoglobin values are within 10 - 12 g/dl | weeks 32-36
  Proportion of subjects with hemoglobin values are within 10 - 12 g/dl for the last 4 weeks of the period for assessment of treatment of efficacy and safety (weeks 32-36)
Incidence of blood transfusions | 52 weak
  Incidence of blood transfusions

OTHER OUTCOMES:
Incidence and nature of adverse events | 52 weak
  Incidence and nature of adverse events
Incidence of drug related adverse events | 52 weak
  Incidence of drug related adverse events
Number of subjects who prematurely withdrew from the study due to AE and SAE | 52 weak
  Number of subjects who prematurely withdrew from the study due to AE and SAE
Number of subjects with presence of anti-erythropoietin antibodies (anti-EPO Ab) | 52 weak
  Number of subjects with presence of anti-erythropoietin antibodies (anti-EPO Ab)

CONTACTS AND LOCATIONS:
Overall Officials: Bolong Miao, Doctoral, Study Director — Shenyang Sunshine Pharmaceutical Co., LTD.
Locations (19):
- Russia (11):
  - State Budgetary Healthcare Institution "Volgogradskiy Regional Center of Urology and Nephrology", Volzhsky, Volgograd Oblast
  - State budgetary healthcare institution of Moscow region "Moscow Regional Scientific Research and Clinical Institute named after M.F.Vladimirsky", Department of Transplantation, nephrology and surgical hemocorrection, Moscow
  - State Budgetary Healthcare Institution of the Republic of Karelia "V.A. Baranov Republican Hospital", Moscow
  - State budgetary healthcare institution "City Clinical Hospital № 1" of Orenburg, Orenburg
  - State Budgetary Educational Institution of Higher Professional Education "North-Western State Medical University named after I.I. Mechnikov " Ministry of Health of Russian Federation, Saint Petersburg
  - The Federal State Budgetary Institute "The Nikiforov Russian Center of Emergency and Radiation Medicine" of the Ministry of Russian Federation for Civil Defense, Emergencies and Elimination of Consequences of Natural Disasters, Saint Petersburg
  - St- Petersburg state budgetary healthcare institution "City Mariinsky Hospital", department of hemodialysis, Saint Petersburg
  - State budgetary institution "St-Petersburg' scientific-research institution of emergency n.a Dzanelidze)", Saint Petersburg
  - St-Peterburg State healthcare institution "Municipal hospital of "Elizabethan Hospital, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Hospital No. 15", Saint Petersburg
  - Federal State Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara
- Thailand (8):
  - Bamrasnaradura Infectious Disease Institute, Bangkok
  - Bhumibol Adulyadej hospital, Bangkok
  - BMA hospital, Bangkok
  - Chulalongkorn King Memorial hospital, Bangkok
  - Klongton Hospital, Bangkok
  - Phramongkutklao hospital, Bangkok
  - Rajavithi hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miao B, Isachkina AN, Shutov EV, Selyutin AA, Kvitkova LV, Shilo VY, Vetchinnikova ON, Alexandrov IV, Perlin DV, Zuev AV, Davydkin IL, Mironova TP, Solovyova OM, Tutin AP, Omelchenko AM, Vareesangthip K, Khadikova NG, Li M, Li X. Biosimilar erythropoietin in anemia treatment (BEAT)-Efficacy and safety of a 1:1 dose conversion from EPREX(R) to EPIAO(R) in patients with end-stage renal disease on hemodialysis: A prospective, randomized, double blind, parallel group study. Medicine (Baltimore). 2022 Nov 25;101(47):e31426. doi: 10.1097/MD.0000000000031426. PMID 36451454

DOCUMENTS (1):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02947438/Prot_000.pdf